CLINICAL TRIAL: NCT01805076
Title: Effect of Preoperative Breast MRI on Surgical Outcomes, Costs and Quality of Life of Women With Breast Cancer
Brief Title: MRI and Mammography Before Surgery in Patients With Stage I-II Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American College of Radiology Imaging Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A011104; ACRIN 6694; U10CA037447 (NIH); NCI-2012-02045 (Registry Identifier: Clinical Trial Reporting Program)
Record Dates: First submitted 2013-02-24; First posted 2013-03-06 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Estrogen Receptor-negative Breast Cancer; Progesterone Receptor-negative Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Mastectomy, Segmental; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (control) (Other): Patients undergo a clinical breast examination and mammography with ultrasound of the breast and regional nodes followed by breast conserving surgery.
  Interventions: Procedure: Breast surgery; Procedure: Mammography
- Arm 2 (experimental) (Experimental): Patients undergo a clinical breast examination, mammography with ultrasound of breast and regional nodes and breast MRI followed by breast conserving surgery or mastectomy.
  Interventions: Procedure: Breast surgery; Procedure: Magnetic resonance imaging; Procedure: Mammography

INTERVENTIONS:
Procedure: Breast surgery
Procedure: Magnetic resonance imaging
  Arms: Arm 2 (experimental)
Procedure: Mammography

SUMMARY:
The purpose of this study is to test whether patients undergoing a breast MRI (magnetic resonance imaging) before breast surgery will have better results after the surgery. Breast tumors are routinely evaluated using mammograms and ultrasound before surgery. This study would like to find out if using MRI in addition to mammography before surgery improves our ability to evaluate tumors and decide what kind of surgery is best for the patient.

DETAILED DESCRIPTION:
This is a randomized trial of preoperative breast MRI in patients deemed eligible for breast conserving surgery by conventional clinical criteria will provide important information about the clinical and biologic relevance of occult disease identified by MRI alone. Patients will be assigned to standard pre-operative breast cancer disease assessment without the addition of MRI prior to breast conserving surgery or standard pre-operative breast cancer disease assessment with the use of MRI prior to breast conserving surgery.

The primary objective is to compare the rates of local-regional recurrence (LRR) following attempted breast conserving therapy in a cohort of women with triple negative or HER-2 amplified breast cancer randomized to preoperative staging with mammography (control arm) or mammography plus breast MRI (MRI arm).

Secondary objectives are:

* To compare the re-operation rates following attempted breast conserving therapy between women assessed preoperatively with breast MRI to those assessed without the use of breast MRI
* To compare local recurrence rates between women who undergo BCT on the control arm to women who undergo BCT on the MRI arm
* To compare the conversion rate to mastectomy secondary to persistent positive margins or poor cosmesis within the first 6 months of attempting BCT (prior to the administration of RT) between women assessed preoperatively with breast MRI to those assessed without the use of breast MRI
* To compare the contralateral breast cancer rates in women randomized to preoperative breast MRI to those not receiving pre-operative breast MRI
* To compare the disease-free survival rates between women assessed preoperatively with breast MRI to those assessed without the use of breast MRI
* To compare breast cancer specific and overall survival outcomes of women assessed preoperatively with breast MRI to those assessed without the use of breast MRI
* To estimate the rate of MRI-guided localization assisted surgery
* To estimate the rate of multi-centric disease in the index breast for women in the MRI arm
* To evaluate the accuracy of index lesion characteristics and other factors in predicting multi-centricity in the cohort randomized to breast MRI
* To assess the positive predictive values (PPV) of MRI in detecting ipsilateral multi-centric disease and contralateral disease in women with breast cancer undergoing preoperative breast MRI
* To estimate the false positive rate for detection of multiple foci of breast cancer by MRI

All registered patients will be monitored for relapse and survival for 5 years from the date of surgery. Patients will be followed a minimum of every 4 months for the first 2 years from diagnosis and a minimum of every 6 months during years 3-5. Patients will be monitored for local, regional, distant relapse and vital status.

ELIGIBILITY:
* Female. Men are excluded from this study because the number of men with breast cancer is insufficient to provide a statistical basis for assessment of effects in this subpopulation of people with breast cancer.
* Pathologically confirmed diagnosis of breast cancer, clinical stage I-II (T1-3 N0 M0, T0-2 N1 M0). Diagnosis must be by needle biopsy; patients diagnosed by surgical excision are excluded.
* Patients must have either:

  * Estrogen receptor (ER) negative/progesterone receptor (PR) negative (< 10% by immunohistochemistry IHC staining) and HER-2 negative breast cancer OR
  * ER negative/PR negative (< 10% by IHC staining) and HER-2 positive tumors
  * HER-2 status will be determined as per the 2013 ASCO CAP guidelines:

    * HER-2 is considered positive if there is IHC 3+ staining or ISH positive using either single probe ISH or dual probe ISH
    * HER-2 is considered negative if there is IHC 0 or 1+ staining or ISH negative using either single probe ISH or dual probe ISH
* No patients with previous ipsilateral invasive breast cancer or ductal carcinoma in situ (DCIS)
* No patients with bilateral breast cancer
* No patients with known deleterious mutations in breast cancer (BRCA) genes
* No current history of receiving hormonal therapy, tamoxifen, and or aromatase inhibitors for therapeutic measures
* No history of chemotherapy for cancer within 6 months prior to registration
* No patients scheduled to receive neoadjuvant chemotherapy or partial breast irradiation following breast conserving surgery
* Eligible for BCT based on clinical examination, mammography and, if standard practice at a given institution, ultrasound and/or tomogram. Women who cannot be appropriately selected for BCT based on these standard imaging studies, and for whom additional imaging is recommended to clarify local disease extent, will not be eligible for this trial.
* No patients with multicentric or multifocal disease scheduled to undergo multiple lumpectomies. Multifocal disease that can be encompassed in a single operative bed can be enrolled.
* Suitable to undergo MRI and receive the contrast agent gadolinium (exclusions follow):

  * No history of untreatable claustrophobia
  * No presence of metallic objects or implanted medical devices in body (i.e., cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
  * No history of sickle cell disease
  * No contraindication to intravenous contrast administration
  * No known allergy-like reaction to gadolinium or moderate or severe allergic reactions to one or more allergens as defined by the American College of Radiology (ACR); patient may be eligible if willing to undergo pre-treatment as defined by the institution's policy and/or ACR guidance
  * No findings consistent with renal failure, as determined by glomerular filtration rate (GFR) < 30 mL/min/1.73 m^2 based on a creatinine level obtained within 28 days prior to registration
  * Weight lower than that allowable by the MRI table
* No prior MRI of study breast within the 12 months prior to registration
* Non-pregnant and non-lactating. Patients of child-bearing potential must have a negative pregnancy test within 7 days prior to registration. Perimenopausal patients must be amenorrheic > 12 months to be considered not of child-bearing potential
* ≥ 18 years of age
* Signed study-specific informed consent prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Local-regional recurrence (LRR) | Up to 5 years

SECONDARY OUTCOMES:
Re-operation rate | Up to 5 years
Conversion rate to mastectomy secondary to persistent positive margins or poor cosmesis | Within the first 6 months
Time to contralateral breast cancer | Up to 5 years post-randomization
Disease-free survival (DFS) | Up to 5 years post-randomization
Overall survival | Up to 5 years post-randomization
Breast cancer specific survival will be measured | Up to 5 years post-randomization
Rate of MRI-guided localization assisted surgery (Arm B) | Up to 5 years
False positive rate for MRI detection of multiple disease foci | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Bedrosian, MD, Study Chair — M.D. Anderson Cancer Center
Locations (179):
- United States (179):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Enloe Medical Center, Chico, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Dekalb Medical Center, Decatur, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Holy Redeemer Hospital and Medical Center, Meadowbrook, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Fox Valley Surgical Associates Limited, Appleton, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Surgical Associates of Neenah SC, Neenah, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin